CLINICAL TRIAL: NCT02614950
Title: Viral Suppression After Analytic Treatment Interruption in Thai Patients Who Initiated Highly Active Antiretroviral Therapy During Acute HIV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SEARCH Research Foundation (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); US Military HIV Research Program (Network)
Responsible Party: Principal Investigator, Nittaya Phanuphak, MD, PhD, Nittaya Phanuphak, MD, PhD, SEARCH Research Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEARCH 022
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Acute HIV Infection; Antiretroviral Treatment Interruption
MeSH Terms: interventions — Treatment Interruption

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment interuption (Experimental)
  Interventions: Other: Treatment interruption

INTERVENTIONS:
Other: Treatment interruption

SUMMARY:
This is a Phase 2, two-step, open-label study of the outcome of analytic treatment interruption (ATI) on patients who started antiretroviral therapy (ART) during Fiebig Stage I of acute HIV infection (AHI), defined as detectable HIV-RNA without detectable p24 antigen or HIV IgM. The primary endpoint will be rate of sustained viral suppression, defined as HIV-1 RNA < 50 cps/ml at 24 weeks after treatment interruption. During ATI subjects will be monitored closely for safety and will have ART re-initiated if they meet predefined clinical, virological, or immunological criteria. In step I, there will be 8 subjects who undergo ATI. An interim analysis for safety will be conducted after 12 weeks. If none of the subjects maintain viral suppression at 12 weeks then no further subjects will be enrolled into the study. If at least 1 out of 8 subjects maintains viral suppression at 12 weeks then an additional 7 subjects will be enrolled in step 2.

At ATI all antiretroviral drugs will be discontinued. Subjects will be monitored with clinical exam, immunological (CD4), and virological (HIV-RNA) testing at baseline and then on a fixed schedule for 24 weeks. ART will be re-initiated immediately if subjects meet any pre-defined clinical, immunological or virological safety endpoints during the monitoring period.

DETAILED DESCRIPTION:
This is a two step open label study of ATI in patients who initiated ART in the earliest detectable stage (Fiebig I) of HIV infection. In step I, eight subjects will discontinue ART for a period of up to 24 weeks. An interim assessment will be conducted after all eight

subjects in step I complete follow-up for 12 weeks. If at least one out of eight subjects maintains viral suppression (HIV-1 RNA < 50 copies/ml) at 12 weeks, then the study will proceed to step 2, in which 7 additional subjects (maximum total sample size of 15) will undergo ATI. The primary endpoint is proportion of subjects who maintain viral suppression at 24 weeks post ATI. Subjects will be monitored frequently for disease progression using clinical, immunological and virological criteria. ART will be re-initiated immediately for any subjects who meet pre-defined criteria for disease progression.

Parent Study Cohort

This is a sub-study of the protocol "Establish and characterize an acute HIV infection cohort in a high-risk population" (SEARCH 010, RV254, WRAIR 1494) implemented at the Thai Red Cross AIDS Research Center in Bangkok, Thailand. From April 2009 through February 2014 the cohort had enrolled 150 patients with acute infection and 145 (97%) are still in active follow-up. All patients in the cohort are offered ART at the time of enrollment through a separately funded protocol; all 145 subjects (100%) in active follow-up are currently on ART. The median age (range) of the cohort is 28 (18-57) years and 90% are men who have sex with men (MSM).

The cohort currently has 50 volunteers who started ART during Fiebig Stage 1, of whom 24 have been on ART for > 24 months and have HIV-1 < 50 copies/ml. Another 13 volunteers have been on ART 6-24 months with undetectable HIV-1 RNA.

During the period of co-enrollment in this substudy, no additional biological specimens will be collected as part of the RV254/SEARCH 010 protocol. Data and samples from this substudy will be shared with the parent protocol.

Criteria to reinitiate ART after ATI

The criteria to restart ART after ATI are designed to protect the subjects from any possible clinical, immunological, or virological adverse effects in the event that their VL rebounds while off ART. The viral load (VL) criterion of > 1,000 copies/ml was chosen because clinical symptoms of HIV infection or significant decline in CD4 count would not be expected at this low level of viremia. The Fiebig I patients in the SEARCH 010 cohort had a median (range) HIV-1 RNA of 4.8 (2.8-5.7) log10copies/ml, at a median (range) of 12 (4-40) days after exposure to HIV, prior to initiation ART and have therefore already been exposed to high levels of plasma virus during acute infection while maintaining low or no detectable HIV proviral reservoirs.

In addition, the ANRS Visconti study found that patients who are virologic controllers (sustained VL < 50 copies/ml) after ATI may initially and transiently have VL above detection. Of 240 tests performed after treatment interruption in those who were subsequently virologic controllers or PTC, 2% had VL > 400 copies/ml and 18% had VL between 50 and 400 copies/ml. Therefore, low-level viremia may not always be indicative of viral rebound and can potentially reverse.

Specific criteria for re-initiation of ART after ATI are:

1. HIV-1 RNA above 1,000 copies/ml on 2 consecutive determinations at least 3 days apart. OR
2. HIV-1 RNA rise of ≥ 0.5 log10copies/ml per day provided that the last HIV-1 RNA is above 1000 copies/ml OR
3. A single HIV-1 RNA above 10,000 copies/ml OR
4. CD4+ T-cell counts below 350 cells/mm3 on 2 consecutive determinations at least 2 weeks apart. OR
5. CD4+ T-cell count decline of > 50% from baseline prior to ATI. OR
6. Clinical progression to CDC Category B or C disease. OR
7. Diagnosis of Acute Retroviral Syndrome. OR
8. Pregnancy OR
9. Subject requests re-initiation of ART.

ELIGIBILITY:
Inclusion Criteria:

* Subject currently enrolled in SEARCH 010/RV254 Acute HIV Infection cohort.
* Male and females aged > 18 years.
* Fiebig Stage I at entry to SEARCH 010/RV254 cohort.
* Taking ART > 24 months.
* HIV-1 RNA < 50 cps/ml for the past 12 months
* Integrated HIV in PBMCs below level of detection (1 copy/105 PBMCs) within the last 6 months
* Most recent (within 3 months) peripheral blood CD4 count > 400 cells/mm3
* No HIV-related or AIDS Defining illness within the last 6 months (Appendix 1)
* Ability and willingness to provide written informed consent.
* Female-specific Criteria:
* Agrees not to become pregnant from the time of study enrollment until the last study visit. If a woman is sexually active and has no history of hysterectomy or tubal ligation or menopause, she must agree to use a prescription birth control method or a barrier birth control method.
* Negative β-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment for any women unless she is post-menopause for 24 consecutive months or has undergone a surgical procedure that precludes pregnancy

Exclusion Criteria:

* Pregnancy or breast-feeding.
* Untreated Syphilis
* Hepatitis B surface antigen positive at any time in the past.
* Hepatitis C antibody positive at any time in the past.
* Serious medical or psychiatric illness that, in the opinion of the site investigator, would interfere with the ability to adhere to study requirements or to give informed consent.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements or to give informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
HIV-1 RNA< 50 cps/ml | 24 weeks after ATI

CONTACTS AND LOCATIONS:
Overall Officials: Nittaya - Phanuphak, MD, PhD, Principal Investigator — SEARCH Research Foundation
Locations (1):
- SEARCH Thailand, Bangkok, Bangkok, Thailand